CLINICAL TRIAL: NCT04814316
Title: Evaluation of the Effects of Lansoprazole Usage on Bone Turnover Markers in Children With Gastroesophageal Reflux or Gastroesophageal Reflux Disease
Brief Title: Effects of Lansoprazole on Bone Turnover Markers
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Islek, Associate Professor, Ataturk University
Other Study IDs: B.30.2.ATA.0.01.00/500
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Bone Turnover Rate Disorder; Calcium Metabolism Disorders
Keywords: Lansoprazole; Bone turnover; Gastroesophageal reflux
MeSH Terms: conditions — Calcium Metabolism Disorders; Gastroesophageal Reflux | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 5ml EDTA blood and 3 ml urine specimens will be collected for each case.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients with gastroesophageal reflux or gastroesophageal reflux disease who will use lansoprazole.
  Interventions: Diagnostic Test: Blood and urine specimens
- Control group: Healty volunteers who will not use lansoprazole.
  Interventions: Diagnostic Test: Blood and urine specimens

INTERVENTIONS:
Diagnostic Test: Blood and urine specimens — Blood and urine samples will be taken at baseline and at the end of the second month. For this purpose, 5 ml of blood samples will be taken to plain blood tubes for evaluation of calcium, magnesium, alkaline phosphatase, parathormone, 25-OH vitamin D and osteocalcin quantities. And 3 ml of urine for calcium, creatinine, deoxypyridinoline, C-terminal telopeptides type-1 collagen and N- terminal telopeptides type-1 collagen.

SUMMARY:
Use of proton pump inhibitors (PPI) has increased in recent years. There are concerns that PPIs have possible negative effects on bone metabolism. It has been suggested that PPIs may reduce the absorption of calcium from the small intestine and lead to bone resorption by affecting osteoclastic activity. In this study, it is planned to investigate the effects of lansoprazole, a proton pump inhibitor, on bone turnover markers in pediatric patients with gastroesophageal reflux or gastroesophageal reflux disease.

DETAILED DESCRIPTION:
This study is planned to be conducted with children who are diagnosed with gastroesophageal reflux or gastroesophageal reflux disease aged 2-18 years and healthy volunteers. The diagnosis of gastroesophageal reflux will be made in accordance with the guidelines of North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition (NASPGHAN) and European Society for Pediatric Gastroenterology, Hepatology, and Nutrition (ESPGHAN). Written and verbal consent will be obtained from patients/healthy volunteers and/or parents who want to participate in the study. Serum calcium, magnesium, alkaline phosphatase, parathormone, 25-OH vitamin D and osteocalcin and urine calcium, creatinine, deoxypyridinoline, C-terminal telopeptides type-1 collagen and N- terminal telopeptides type-1 collagen levels will be measured at baseline and second month in study group and once in control groups.

ELIGIBILITY:
Inclusion Criteria:

• Patients diagnosed with gastroesophageal reflux or gastroesophageal reflux disease aged 16 to18 years.

Exclusion Criteria:

* Patients with a malabsorptive disease.
* Patients with any chronic disease.
* Patients who use any medication that may affect calcium and bone metabolism.
* Patients who used proton pumps inhibitor within the last 3 months.
* Patients who do not use lansoprazole in the study group.
* Patients whose blood and urine samples are not taken in the eighth week of treatment.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with gastroesophageal reflux or gastroesophageal reflux disease aged 16 to18 years who were treated in Pediatric Gastroenterology Department of Ataturk University Hospital included to the study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Measuring serum calcium levels | First day
  Measuring serum calcium levels with spectrophotometric method (mg/dL).
Measuring serum alkaline phosphatase levels | First day
  Measuring serum alkaline phosphatase levels with spectrophotometric method (U/L).
Measuring serum magnesium levels | First day
  Measuring serum magnesium levels with spectrophotometric method (mg/dL).
Measuring serum osteocalcin levels | First day
  Measuring serum osteocalcin levels with spectrophotometric method (mg/L).
Measuring serum parathyroid hormone levels | First day
  Measuring serum parathyroid hormone levels with immunoassay method (pg/mL).
Measuring serum vitamin D levels | First day
  Measuring serum vitamin D with immunoassay method (ng/mL).
Measuring urine deoxypyridinoline levels | First day
  Measuring urine deoxypyridinoline levels with immunoassay method (nmol DPD/mmol creatinine).
Measuring spot urine calcium levels | First day
  Measuring urine calcium levels with spectrophotometric method (mg/dL).
Measuring urine creatinine levels | First day
  Measuring urine creatinine levels with spectrophotometric method (mg/dL).
Measuring urine C-terminal telopeptides Type I collagen levels | First day
  Measuring urine C-terminal telopeptides Type I collagen levels with immunoassay method (ng/mL).
Measuring urine N-terminal telopeptides Type I collagen levels | First day
  Measuring urine N-terminal telopeptides Type I collagen levels with immunoassay method (ng/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Ali Islek, MD, Principal Investigator — Ataturk University School of Medicine
Locations (1):
- Ataturk University Hospital, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sheraly AR, Lickorish D, Sarraf F, Davies JE. Use of gastrointestinal proton pump inhibitors to regulate osteoclast-mediated resorption of calcium phosphate cements in vivo. Curr Drug Deliv. 2009 Apr;6(2):192-8. doi: 10.2174/156720109787846225. PMID 19450226
- [Result] Targownik LE, Lix LM, Metge CJ, Prior HJ, Leung S, Leslie WD. Use of proton pump inhibitors and risk of osteoporosis-related fractures. CMAJ. 2008 Aug 12;179(4):319-26. doi: 10.1503/cmaj.071330. PMID 18695179
- [Result] Yang YX, Lewis JD, Epstein S, Metz DC. Long-term proton pump inhibitor therapy and risk of hip fracture. JAMA. 2006 Dec 27;296(24):2947-53. doi: 10.1001/jama.296.24.2947. PMID 17190895
- [Result] Targownik LE, Lix LM, Leung S, Leslie WD. Proton-pump inhibitor use is not associated with osteoporosis or accelerated bone mineral density loss. Gastroenterology. 2010 Mar;138(3):896-904. doi: 10.1053/j.gastro.2009.11.014. Epub 2009 Nov 18. PMID 19931262
- [Result] Sharara AI, El-Halabi MM, Ghaith OA, Habib RH, Mansour NM, Malli A, El Hajj-Fuleihan G. Proton pump inhibitors have no measurable effect on calcium and bone metabolism in healthy young males: a prospective matched controlled study. Metabolism. 2013 Apr;62(4):518-26. doi: 10.1016/j.metabol.2012.09.011. Epub 2012 Oct 24. PMID 23102518
- [Result] Kocsis I, Arato A, Bodanszky H, Szonyi L, Szabo A, Tulassay T, Vasarhelyi B. Short-term omeprazole treatment does not influence biochemical parameters of bone turnover in children. Calcif Tissue Int. 2002 Aug;71(2):129-32. doi: 10.1007/s00223-001-2068-9. Epub 2002 Jul 23. PMID 12200646
- [Result] Qvist P, Christgau S, Pedersen BJ, Schlemmer A, Christiansen C. Circadian variation in the serum concentration of C-terminal telopeptide of type I collagen (serum CTx): effects of gender, age, menopausal status, posture, daylight, serum cortisol, and fasting. Bone. 2002 Jul;31(1):57-61. doi: 10.1016/s8756-3282(02)00791-3. PMID 12110413